CLINICAL TRIAL: NCT01440088
Title: A Randomized Phase 3, Multicenter, Open-Label Study Comparing TH-302 in Combination With Doxorubicin vs. Doxorubicin Alone in Subjects With Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma
Brief Title: A Trial of TH-302 in Combination With Doxorubicin Versus Doxorubicin Alone to Treat Patients With Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Collaborators: Sarcoma Alliance for Research through Collaboration (SARC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-406/SARC021
Expanded Access: NCT02712567 (No longer available)
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: TH-302; TH-CR-406; SARC021; Locally Advanced Soft Tissue Sarcoma; Metastatic Soft Tissue Sarcoma; Sarcoma; Doxorubicin; Evofosfamide
MeSH Terms: conditions — Sarcoma | interventions — TH 302; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TH-302 in Combination with Doxorubicin (Experimental)
  Interventions: Drug: TH-302 in Combination with Doxorubicin
- Doxorubicin (Active Comparator)
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: TH-302 in Combination with Doxorubicin — 300 mg/m2 of TH-302 will be administered by IV infusion over 30-60 minutes on Days 1 and 8 of a 21-day cycle.
  Doxorubicin may be delivered as a bolus administration or as a continuous infusion administration; administration schedule must be specified prior to enrollment.
  Doxorubicin bolus administration: 75 mg/m2 administered by bolus injection starting on Day 1 of a 21-day cycle.
  Doxorubicin continuous administration: 75 mg/m2 administered by continuous IV infusion over 48-96 hours starting on Day 1 of a 21-day cycle.
  Doxorubicin administration will start between 2 to 4 hours after completion of the TH-302 infusion when used in combination with TH-302.
  Arms: TH-302 in Combination with Doxorubicin
Drug: Doxorubicin — Doxorubicin may be delivered as a bolus administration or as a continuous infusion administration; administration schedule must be specified prior to enrollment.
  Doxorubicin bolus administration: 75 mg/m2 administered by bolus injection starting on Day 1 of a 21-day cycle.
  Doxorubicin continuous administration: 75 mg/m2 administered by continuous IV infusion over 48-96 hours starting on Day 1 of a 21-day cycle.
  Arms: Doxorubicin

SUMMARY:
The purpose of this study is to determine whether TH-302 in combination with Doxorubicin is safe and effective in the treatment of Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma.

DETAILED DESCRIPTION:
TH-302 is designed to target the hypoxic regions of tumors which are generally located distant from tumor vessels. Doxorubicin has poor tissue penetration and targets the regions of tumors that are located in proximity to the tumor vessels. The presence of hypoxia in solid tumors is associated with a more malignant phenotype and resistance to chemotherapy. The hypoxia-activated prodrug, TH-302, is designed to selectively target the hypoxic microenvironment. Soft tissue sarcomas have evidence supporting the presence of hypoxia based on pO2 histography, F-MISO and gene expression profiling. There is an absence of therapeutic options for subjects with soft tissue sarcoma. Combining doxorubicin with TH-302 may enable the targeting of both the normoxic and hypoxic regions of soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 15 years of age
* Ability to understand the purposes and risks of the study and has signed or, if appropriate, the subject's parent or legal guardian has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Pathologically confirmed diagnosis of soft tissue sarcoma of the following histopathologic types:

  * Synovial sarcoma
  * High grade fibrosarcoma
  * Undifferentiated sarcoma; sarcoma not otherwise specified (NOS)
  * Liposarcoma
  * Leiomyosarcoma (excluding GIST)
  * Angiosarcoma (excluding Kaposi's sarcoma)
  * Malignant peripheral nerve sheath tumor
  * Pleomorphic Rhabdomyosarcoma
  * Myxofibrosarcoma
  * Epithelioid sarcoma
  * Undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma (MFH) (including pleomorphic, giant cell, myxoid and inflammatory forms)
* Locally advanced unresectable or metastatic disease with no standard curative therapy available and for whom treatment with single agent doxorubicin is considered appropriate.
* Recovered from reversible toxicities of prior therapy
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Acceptable liver, renal, hematological and cardiac function
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception

Exclusion Criteria:

* Prior systemic therapy for advanced or metastatic disease (neoadjuvant therapy followed by surgical resection and adjuvant therapy permitted). Palliative radiotherapy to non-target lesions is allowed if completed at least two weeks prior to study entry
* Low grade tumors according to standard grading systems
* Prior therapy with ifosfamide or cyclophosphamide or other nitrogen mustards
* Prior therapy with an anthracycline or anthracenedione
* Prior mediastinal/cardiac radiotherapy
* Current use of drugs with known cardiotoxicity or known interactions with doxorubicin
* Anti-cancer treatment with radiation therapy, neoadjuvant or adjuvant chemotherapy, targeted therapies, immunotherapy, hormones or other antitumor therapies within 4 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C). Palliative radiotherapy to non-target lesions is allowed, is completed at least two weeks prior to study entry.
* Significant cardiac dysfunction precluding treatment with doxorubicin
* Seizure disorders requiring anticonvulsant therapy unless seizure-free for the last year
* Known brain metastases (unless previously treated and well controlled for a period of ≥ 3 months)
* Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
* Severe chronic obstructive or other pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Prior therapy with a hypoxic cytotoxin
* Subjects who participated in an investigational drug or device study within 28 days prior to study entry
* Known infection with HIV, hepatitis B, or hepatitis C
* Subjects who have exhibited allergic reactions to a structural compound similar to TH-302,doxorubicin or their excipients
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of TH-302 in combination with doxorubicin | 2 years
  Efficacy will be determined by overall survival in subjects with locally advanced unresectable or metastatic soft tissue sarcoma previously untreated with chemotherapy compared with doxorubicin alone

SECONDARY OUTCOMES:
Safety of TH-302 in combination with doxorubicin in subjects with locally advanced unresectable or metastatic soft tissue sarcoma compared with doxorubicin alone | 2 years
  To investigate the pharmacokinetics of TH-302, Br-IPM, doxorubicin, and doxorubicinol in plasma

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (92):
- United States (44):
  - Mayo Arizona, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - USC-Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - South Florida Center for Gynecologic Oncology, Boca Raton, Florida
  - Mayo Clinic-Florida-Cancer Clinical Studies Unit, Jacksonville, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - H.Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Midtown Campus, Atlanta, Georgia
  - Kootenai Health - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Health Care - University of Iowa Hospital, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute Center for Sarcoma and Bone Oncology, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Mayo Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore, The Bronx, New York
  - Carolinas Hematology-oncology Associates-Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Arthur G. James Cancer Hospital and Richard J Solove Research Institue, The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - MUSC - Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth Universtiy-Massey Cancer Center, Richmond, Virginia
  - University of Washington Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (3):
  - University Klinikum Graz, Graz
  - Univ. Klinik fur Innere Medizin I Internistische Onkologie Medizinische Universitat Innsbruck, Innsbruck
  - Allgemeines Krankenhaus Wien, Vienna
- Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg, Leuven, Belgium
- Canada (7):
  - Juravinski Cancer Centre at Hamilton Health Sciences - Department of Medicine, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Tom Baker Cancer Centre, Calgary
  - Cross Cancer Institute, Edmonton
  - Ottawa Health Research Institue, Ottawa
  - BCCA- Vancouver Cancer Centre - Division of Medical Oncology, Vancouver
  - Cancer Care Manitoba, Winnipeg
- University Hospital Herlev at Copenhagen, Herlev, Copenhagen, Denmark
- France (8):
  - ICO Rene Gauducheau, Saint-Herblain, Nantes
  - Institut Bergonie, Bordeaux
  - Departement d'Oncologie Medicale, Dijon
  - Centre Leon Berard, Lyon
  - Département d'Oncologie Moléculaire, Institut Paoli-Calmettes (IPC) and U119 Inserm, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
- Germany (7):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Helios Klinikum Bad Saarow, Department of Hematology, Oncology, and Palliative Care, Sarcoma Center Berlin-Brandenburg, Berlin
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Medizinische Hochschule Hannover (MHH) - Klinik fuer Haemonstaseologie, Onkologie und Stammzelltransplantation, Hanover
  - Div. of Surgical Oncology & Thoracic Surgery, Mannheim University Medical Center, Mannheim
  - Wilhelm's University, Universitatsklinikum Muenster, Medizinische Klinik und Poliklinik A, Albert-Schweitzer-Campus 1, Münster
- Hungary (2):
  - Magyar Honvedseg Honvedkorhaz, Onkologiai Osztaly, Budapest
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Megyei Onkologiai Kozpont, Szolnok
- Sharette Institute of Oncology, Hadassah-Hebrew University Medical Center, Hadassah Medical Org-Ein Karem, Kiryat Hadassah, Jerusalem, Israel
- Italy (6):
  - IRCCS Centro di Riferimento Oncologico-Struttura Operativa, Aviano, Pordenone
  - Fondazione del Piemonte per l'Oncologia, Instituto per la Ricerca e la Cura del cancro (I.R.C.C.), Dipartimento Oncologico, Direzione Operativa Oncologia Medica a Direzione Universitaria, Candiolo, Torino
  - Centro di Riferimento Oncologico (CRO), Aviano
  - Azienda Ospedaliera Garibaldi, Catania
  - Azienda Ospedaliero Universitaria-Policlinico Paolo Giacco, Palermo
  - ASL TO/2 di TORINO_Presidio Sanitario Gradenigo, S.C. di Oncologia, Torino
- Poland (3):
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Centrum Onkologii Instytut im M. Sklodowskiej-Curie, Krakow
  - Centrum Onkologii-Instytut im. M. Sklodowskiej-Curie, Warsaw
- Russia (3):
  - GUZ "Regional Oncology Dispensay", Kazan, Kazan'
  - ROTSN RAMS them. Н.Н.Блохина NN Blokhin, Moscow
  - FGU Moscow Research Institute of Oncology named after P.A. Hertzen of Rosmedtechnology, Moscow
- Spain (6):
  - H.U. Canarias, Hospital Universitario de Canarias. Servicio de Oncología Médica, Santa Cruz de Tenerife, Canary Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Sant Joan de Deu, Department de Oncologia, Barcelona
  - Hospital Universitario Ramón y Cajal., Madrid
  - Universidad Complutense Madrid Facultad de Medicina - Hospital Universitario 12 de Octubre, Servicio de Oncologia Medica Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Derived] Tap WD, Papai Z, Van Tine BA, Attia S, Ganjoo KN, Jones RL, Schuetze S, Reed D, Chawla SP, Riedel RF, Krarup-Hansen A, Toulmonde M, Ray-Coquard I, Hohenberger P, Grignani G, Cranmer LD, Okuno S, Agulnik M, Read W, Ryan CW, Alcindor T, Del Muro XFG, Budd GT, Tawbi H, Pearce T, Kroll S, Reinke DK, Schoffski P. Doxorubicin plus evofosfamide versus doxorubicin alone in locally advanced, unresectable or metastatic soft-tissue sarcoma (TH CR-406/SARC021): an international, multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1089-1103. doi: 10.1016/S1470-2045(17)30381-9. Epub 2017 Jun 23. PMID 28651927
- [Derived] Chawla SP, Cranmer LD, Van Tine BA, Reed DR, Okuno SH, Butrynski JE, Adkins DR, Hendifar AE, Kroll S, Ganjoo KN. Phase II study of the safety and antitumor activity of the hypoxia-activated prodrug TH-302 in combination with doxorubicin in patients with advanced soft tissue sarcoma. J Clin Oncol. 2014 Oct 10;32(29):3299-306. doi: 10.1200/JCO.2013.54.3660. Epub 2014 Sep 2. PMID 25185097